CLINICAL TRIAL: NCT00346593
Title: Investigation of the Clinical Performance of Silicone Hydrogel Contact Lenses During Continuous Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Clinical Vision Research Australia (Other); Cooper Companies (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H03 010
Record Dates: First submitted 2006-06-29; First posted 2006-06-30 (Estimated); Last update posted 2007-02-12 (Estimated); Status verified 2007-02

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

INTERVENTIONS:
Device: Silicone hydrogel contact lens

SUMMARY:
The primary purpose of this study is to investigate the clinical performance of a new silicone hydrogel contact lens during continuous wear (up to 30 nights) over a period of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Has had an oculo-visual examination in the last 2 years.
* Is correctable to at least 6/7.5 distance visual acuity in each eye with spherical contact lenses.
* Is a current soft contact lens wearer.
* Has no clinically significant anterior eye findings.
* Has no other active ocular disease.

Exclusion Criteria:

* Has any systemic disease that might interfere with contact lens wear
* Is using any systemic or topical medications that will affect ocular health.
* Has any pre-existing ocular irritation that would preclude contact lens fitting.
* Has any ocular pathology or severe insufficiency of lacrimal secretion (dry eyes) that would affect the wearing of contact lenses.
* Has undergone corneal refractive surgery.
* Is pregnant, lactating or planning a pregnancy.

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Dates: Start 2004-05; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Carol Lakkis, BScOptom PhD, Principal Investigator — Clinical Vision Research Australia
Locations (1):
- Clinical Vision Research Australia, Carlton, Victoria, Australia